CLINICAL TRIAL: NCT06632132
Title: Boosting Knowledge, Attitudes, and Practices: An Experimental Study Evaluating the Effectiveness of mHealth Training on Antimicrobial Resistance for Hemodialysis Nurses
Brief Title: Antimicrobial Resistance Training for Hemodialysis Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/581
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Antimicrobial Resistance in Hemodialysis
Keywords: Antimicrobial Resistance; Hemodialysis Unit; mhealth; Chatbot; Knowledge; Practice; Attitudes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis nurses receiving antimicrobial resistance training (Experimental): Hemodialysis nurses received educational program about antimicrobial resistance and uses in hemodialysis units. The program developed by the researcher is meticulously designed, drawing on extensive insights from the WHO curricula guide (nurses' education and training on antimicrobial resistance; 2019) and the literature review addressed the use of antibiotics and prevention of AMR in hemodialysis facilities.
  Interventions: Other: Antimicrobial resistance Training in Hemodialysis Units
- Control group (No Intervention): they were no given any educational content about the study intervention during the study. However, they were provided with the educational material received by experimental group via Chatbot software after evaluation completed

INTERVENTIONS:
Other: Antimicrobial resistance Training in Hemodialysis Units — The educational program developed by the researcher is meticulously designed, drawing on extensive insights from the WHO curricula guide (nurses' education and training on antimicrobial resistance; 2019) and the literature review addressed the use of antibiotics and prevention of AMR in hemodialysis facilities. The curriculum, using simple English, provides a broad set of learning objectives tailored to the expected roles of nurses.
  The education program includes four main modular outline:
  1. Foundations that build awareness of antimicrobial resistance
  2. Appropriate use of antimicrobial agents
  3. Infection prevention and control
  4. Diagnostic stewardship and surveillance
  The educational material was sent by a study researcher (X) to the WhatsApp number for all members of the experimental group via Chatbot software, which was designed by software engineer. The educational materials were sent in the form of written materials, photos, and videos.
  Arms: Hemodialysis nurses receiving antimicrobial resistance training

SUMMARY:
Objective: To evaluate the impact of an m-health training program on nurses' knowledge, attitudes, and practices concerning antimicrobial resistance (AMR) within hemodialysis units.

Design: This study utilized a controlled experimental design with cluster random assignment, adhering to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

Method: A convenience sample of 64 nurses was cluster-randomized into either an experimental group (n = 32) or a control group (n = 32). The experimental group received AMR education via WhatsApp using Chabot software, while the control group received the same content through leaflets. The nurses' knowledge, attitudes, and practices regarding AMR were assessed with self-developed instruments at three time points: baseline (Time 1), immediately after the intervention (Time 2), and one month later (Time 3).

DETAILED DESCRIPTION:
Introduction

Patients undergoing hemodialysis treatment are at an increased risk for infections because these patients require prolonged healthcare interventions, have weakened immune system, use antibiotics, receive treatment in a shred healthcare setting, and require vascular accesses such as catheters, fistulas and venous central lines. Infection is the second master cause of mortality in hemodialysis population, accounting for 8% of all deaths. to the general population, hemodialysis patients have higher rates of infection, particularly sepsis and its associated mortality.

Due to the high rate of infections among hemodialysis patients, there is a significant utilization of antimicrobial agents in this population. This extensive use has led to the emergence of multidrug-resistant organisms in hemodialysis units. Antimicrobial resistance (AMR) arises when microorganisms, including bacteria, fungi, viruses, and parasites, evolve mechanisms to resist the effects of antimicrobial agents. In recent years, there has been an increase in the prevalence of AMR in hemodialysis facilities worldwide, particularly among bacteria such as Staphylococcus aureus, Escherichia coli, and Klebsiella pneumonia. Staphylococcus aureus causes up to 70 % of vascular access infections in hemodialysis patients, and the problem worsens by the dissemination of methicillin-resistant S. aureus (MRSA) isolates. About 90 % of patients with MRSA infections require hospitalization, and 17 % die during hospital stay.

In Jordan, gram-positive bacterial infections and antibiotic resistance rates were high in Jordan. Methicillin-resistant S. aureus (MRSA) and methicillin-resistant coagulase-negative Staphylococci (MR-CoNS) infections were common and exhibited high rates of antibiotic resistance. Furthermore, streptococcus pneumonia showed increased resistance rates to most antimicrobials. Reports form Jordanian hospitals also showed a high prevalence of AMR, with particular note to methicillin-resistant Staphylococcus aureus (MRSA) that reached a rate of 45% (Ministry of Health National Action Plan, 2018).

Antimicrobial resistance is a complex and multifaceted global public health issue that threatens the effective prevention and treatment of infections. In 2019, the World Health Organization (WHO) announced AMR as one of the top 10 global public health threats facing humanity in 2019. Antimicrobial resistance renders standard treatments ineffective, complicating infection management, and elevating the risk of disease transmission, prolonged illness, and adverse outcomes. It also leads to increased morbidity, mortality, and hospital stays. The cost of AMR to the economy is significant as well. In addition to death and disability, prolonged illness results in longer hospital stays, leading to more expensive medications and increased financial burdens for those effected. AMR is predicted to cost the world economy between $300 billion and $1 trillion by 2050.

To mitigate the risk of antimicrobial resistance among patients undergoing hemodialysis, it is essential to implement stringent infection prevention and control measures. Additionally, raising awareness among healthcare providers, patients, and caregivers about the importance of responsible antibiotic use and infection prevention is crucial. Nurses play a crucial role in the management of AMR generally and in hemodialysis facilities specifically. They can promote the appropriate use of antimicrobial drugs and implement effective infection prevention and control measures. However, existing literature indicates that nurses often lack knowledge, attitudes, and skills related to various dimensions of antimicrobial resistance (AMR) in hemodialysis patients. This highlights the need for developing and implementing effective and innovative continuous educational programs to address these gaps.

Recently, advanced technology has made it possible to implement new types of behavioral change education. Mobile health (m-Health) is an example. The WHO defines m-Health as medical and public health practice supported by mobile devices, such as mobile phones, patient monitoring devices, personal digital assistants (PDAs), and other wireless devices. By making health information and existing health services more easily and remotely accessible, m-Health technologies are used to improve health and change health behaviors. Short Messaging Service (SMS) and Multimedia Messaging Service (MMS) as common examples of m-health are used to deliver cost-effective health promotion or behavior change interventions, regardless of geography. SMS and MMS require less effort, time, and human resources than phone calls or face-to-face meetings or appointments because they can be sent quickly and easily. Thus, given the ease of use of SMS or MMS, they could be used for potential health behavioral changes or risk reduction with little demand on staff or clinic resources.

Few studies have examined AMR training for nurses. Hendy et al. and Lutfiyati et al. both found that training on antimicrobial stewardship significantly improved nurses' knowledge, attitudes, and practices. Boban et al. observed significant improvement in the antimicrobial resistance knowledge and attitudes in higher education students, including nurses. Similarly, Kpokiri et al. noted that AMR training enhanced overall knowledge of antibiotic use and resistance among healthcare professionals.

Most prior research has focused on traditional training interventions, highlighting a gap in exploring the potential, advantages, and effectiveness of mobile technology for AMR training. Although mobile health applications (MHAs) have been utilized for AMR training in various healthcare settings, their application in hemodialysis units remains unexplored. This identified gap is particularly relevant given the increasing need for mobile technologies to enable continuous education and provide timely cost-effective assistance to health professionals. The current study aimed to address this gap by examining the effectiveness of a mobile health training program on antimicrobial resistance among the knowledge, attitudes, and practices of nurses employed in hemodialysis units.

The results of this study are clinically significant to improve patient care and safety by enhancing practices regarding AMR. Theoretically, it helps facilitate insight on the use of technology for effective health education and behavior change. This research improves the theoretical understanding of the effectiveness of mobile learning platforms by measuring their impact on specific learning outcomes-knowledge, attitudes, and practices-within a specialized health care context. It also adds to the growing body of evidence regarding the role of innovative educational methods in professional development.

Method and Materials Research Design The study employed a pre/posttest randomized controlled experimental design. The study participants were selected using a convenience sampling method and then distributed randomly into the study groups (1:1) by a cluster random assignment, sequence generated by Random Allocation Software, this precaution taken to reduce contamination. The study involved two groups including the experimental and control groups. The experimental group received education about the use of antibiotics and prevention of AMR in HD units using the WhatsApp application via Chatbot software. However, the control group received the same educational content using the leaflets. The details of interventions were explained under the intervention section below.

Sample and Setting

Participants were selected from four major hospitals representing the private, military, public sectors.

The sample size was calculated using the G-power software (Version 3.1.7). With an alpha level of 0.05, a statistical power of 0.9, an effect size of .19 (Alhawatmeh et al., 2022), and a repeated-measures ANOVA test (mixed model), the minimum required total sample size was calculated to be 60 participants. Considering a 15% attrition rate, 9 participants were added, resulting in a final required sample size of 69. Out of the 69 participants initially recruited, 64 completed the study.

Intervention

The educational program developed by the researcher is meticulously designed, drawing on extensive insights from the WHO curricula guide (nurses' education and training on antimicrobial resistance; 2019) and the literature review addressed the use of antibiotics and prevention of AMR in hemodialysis facilities. The curriculum, using simple English, provides a broad set of learning objectives tailored to the expected roles of nurses.

The education program includes four main modular outline:

1. Foundations that build awareness of antimicrobial resistance, which includes the subtopics of Systemic approach to the individual with an infection and Understanding antimicrobial agents and their management.
2. Appropriate use of antimicrobial agents, which include the subtopic of Use of antimicrobial agents in clinical management.
3. Infection prevention and control, which includes the subtopics of Health care-associated infection, antimicrobial resistance and infection prevention and control.
4. Diagnostic stewardship and surveillance, which includes the subtopics of Interaction between diagnostic stewardship and surveillance of antimicrobial resistance and overall antimicrobial stewardship.

For the experimental group, the educational material was sent by a study researcher (X) to the WhatsApp number for all members of the experimental group via Chatbot software, which was designed by software engineer. This software is a strategic move that holds immense potential for transforming the way nurses access information and support. In the dynamic and demanding field of healthcare, nurses often face time constraints and require immediate access to relevant resources. A WhatsApp Chatbot designed for nursing education can serve as a virtual companion, providing real-time assistance and information crucial to their roles. The way information is presented and shared in a Chatbot is one of the most important factors that directly affects the user experience. In contrast to conventional interfaces, a Chatbot method is usually more dynamic and user-friendly since information is frequently communicated through conversational engagements (Fitria et al, 2023). AMR training program was presented in Chatbot software as outlines. The educational materials were sent in the form of written materials, photos, and videos. The study researcher (X) who was an experienced nurse with a master's degree in nursing explained how to use program to each nurse in experimental group by the following instructions and directions:

The program was auto-reply with the educational dialogue that had been previously entered to this program. Also, the researcher advised the participant to read each part carefully. Nurses were able to return to the researchers in order to clarify the vague points and answer any questions via telephone numbers. The application allows the researcher to view the parts that have been accessed and read by participants in the educational program. During one week, nurses in experimental group completed the AMR training program, then the Chabot software was closed before evaluation phase started.

For the control group, they were given the same educational content using leaflets. Nurses in control group were provided with the educational material received by experimental group via Chatbot software after evaluation completed.

Pilot Testing and Content Validity

The tools and educational program were subjected to content validity assessment (CVI) by a panel of four experts in the field of medicine, clinical pharmacology, infection control and nursing. The tool items were overlaid in a matrix with tow option rating scale: 1) Importance which is divided to 3 rating scales (Not necessary, Useful but not necessary, Essential), and 2) relevance that is divided into 4 rating scales (Not relevant/not clear, Item needs some revision, Relevant/ clear but need minor revision, very relevant/clear).

Statistics were subsequently used to assess the degree of reviewers' agreement on the importance and relevance of the tool items. The Content Validity Index values for the Knowledge of Antimicrobial Use and Antimicrobial Resistance, the Attitudes Toward Antimicrobial Use and Antimicrobial Resistance, the practice of Antimicrobial Use and Antimicrobial Resistance were 0.978 0.927 and 0.977 respectively. These values indicated an acceptable level of validity index values.

A pilot study was conducted on 15 registered nurses working in HD units to assess the clarity, objectivity, and feasibility of the study self-developed instruments and the educational programs' content. Through the pilot study, the time required for data collection was estimated. The nurses in the pilot study were not included in the main study sample.

Data Collection Procedure

Institutional Review Board (IRB) approval was obtained prior to commencing the study, followed by securing administrative approvals from the respective study settings. A list of nurses working in the hemodialysis units was then acquired from the head nurse of each unit at the target hospitals. This list included the names and telephone numbers of the nurses. After obtaining the list of nurses, each nurse was contacted by phone. The call followed these steps: the researcher introduced themselves, explained the purpose of the call and the study, and sought verbal consent from the nurse to participate if they met the study criteria. The researcher then gathered information from each nurse to assess their eligibility for the study.

A list of nurses who met the study criteria was compiled, including their work shifts (A, B, and C) and the names of their respective hospitals. We ensured that the nurses in each shift remained in the same shift throughout the duration of the study. Each shift at each hospital was treated as a cluster, with 6 participants recruited from each cluster. This resulted in the identification of 12 clusters (4 hospitals × 3 shifts). These 12 clusters were then randomly assigned to either the experimental or control group using computer-generated randomization, resulting in 6 clusters in each group. This randomization strategy was carried out by an independent researcher who was not involved in the recruitment process and remained blinded to the participant list. The purpose of employing cluster randomization was to prevent contamination between the intervention and control groups.

The researchers scheduled a meeting and interviewed each eligible nurse individually to obtain written consent and implement the baseline measurement. Upon written consent obtained by the study researchers, a well-trained nurse - a research assistant- from each hospital took the nurses' names from the researchers without knowing which of the two groups the nurse was assigned to. A well-trained nurse - a research assistant- from each hospital took the nurses' names from the researcher without knowing which of the two groups the nurse was assigned to. All nurses received the self-administered questionnaire from the research assistants. On the same day, the questionnaires were collected once the nurses had finished. The average time to complete the questionnaire was 30 minutes. The data obtained during this phase served as the baseline (Time 1). The same questionnaire, excluding the demographic characteristics, was completed again by the two study groups immediately at the end of interventions (Time 2) and one month later (Time 3). Each participant completed the study questionnaire individually in a private, quiet room in the hospital without anyone else present, including the research assistant.

Ethical Consideration Ethical approval was obtained from the Institutional Review Board (IRB) (Number: 2023/581). Informed written consent was obtained from participants following a thorough explanation of the study. All data were securely stored in a locked cabinet at the principal investigator's office, and participants' names were replaced with codes to ensure confidentiality. Participants were informed of their right to withdraw from the study at any time.

Data Analysis The Statistical Package for Social Sciences (SPSS version 26) will be used for analyzing the study data. The internal consistency reliability of the study instruments was tested using Cronbach's alpha. Descriptive statistics such as mean, standard deviation, percentage and frequency will be used to describe the study variables. For each main study variable, repeated-measures ANOVA test (within groups) will examine the mean differences over time for each group separately. Also, repeated-measures ANOVA tests (mixed model) will examine the mean score differences between the study groups over time. P-values of 0.05 or less will be used to determine whether the results are statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working at hemodialysis unit
* having smart phones
* ability of reading and writing in English
* commitment to complete all study protocol

Exclusion Criteria:

* Hemodialysis nurses who have taken training about the prevention of AMR and antibiotic uses or the infection control measures in hemodialysis units
* Hemodialysis nurses with less than three months of clinical experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Knowledge of Antimicrobial Use and Resistance | From enrollment to one month post-training completion
  A Self- developed questionnaire to assess the dialysis nurses' knowledge of antimicrobial use and resistance included 28 true and false questions. The answer choices constituting each of the questions were True, False, and I do not know. One point was given for each right answer and 0 points for each wrong answer. If participants selected the choice of "I do not know" for certain question, they would be given 0 on that question. The maximum possible score was 28 points with a range from 0 to 28 points. A higher total score indicated a higher level of knowledge of antimicrobial use and resistance
Attitudes Toward Antimicrobial Use and Resistance | From enrollment to one month post-training completion
  The self-developed scale to measure the dialysis nurses' attitude toward antimicrobial use and resistance includes 11 well-formulated items. Each item was rated on a five-point Likert-type scale (strongly disagree (1) to strongly agree (5)). The maximum possible score was 55 with a range from 11 to 55 points. A higher score means the participants had a more positive attitude toward the appropriate use of antimicrobials and higher sensitivity to antimicrobial resistance
Practice of Antimicrobial Use and Resistance | From enrollment to one month post-training completion
  The self-developed questionnaire to evaluate the dialysis nurses' practice regarding the proper use of antimicrobials and the issue of antimicrobial resistance, includes 27 well-formulated items. Each item was assessed on five-point Likert scale, which ranges from 1 (never) to 5 (always). The total scale ranges from 27 to 135. A higher score of this scale indicated higher strictness of antimicrobial use practices and strong compliance with protocols to prevent antimicrobial resistance

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, Principal Investigator — Hossam alhawatmeh, associate professor, Jordan university of science and technology
Locations (1):
- Prince Rashid Ben AL-Hasan Militarily Hospital under the Jordanian Royal Medical Services (JRMS), Al-Hussein Hospital at King Hussein Medical City, Princess Haya Bent Al-Hussein military hospital, and King Abdullah University Hospital (KAUH)., Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No
Due to ethical constraints, we are unable to share the study data with external parties

REFERENCES:
- [Background] AbuTaha SA, Al-Kharraz T, Belkebir S, Abu Taha A, Zyoud SH. Patterns of microbial resistance in bloodstream infections of hemodialysis patients: a cross-sectional study from Palestine. Sci Rep. 2022 Oct 26;12(1):18003. doi: 10.1038/s41598-022-21979-7. PMID 36289278
- [Background] Al-Tamimi, M., Albalawi, H., Isied, W., Musallam, A., Qazzaz, F., Azab, M., & Abu-raideh, J. (2022). Gram-positive bacterial infections and antibiotics resistance in jordan: current status and future perspective. Jordan Medical Journal, 56(1), Article 1. https://doi.org/10.35516/jmj.v56i1.219.
- [Background] Boban, D., Kaur, K., Greco, S., Pradhan, H. S., Joshi, R., Rakshitha, K., & Prakash, J. (2023). The impact of antibiotic resistance training programs on knowledge, attitude, and practice reflection among Indian higher education students. International Journal of One Health, 87-94. https://doi.org/10.14202/IJOH.2023.87-94.
- [Background] Buhi, E. R., Trudnak, T. E., Martinasek, M. P., Oberne, A. B., Fuhrmann, H. J., & McDermott, R. J. (2013). Mobile phone-based behavioural interventions for health: A systematic review. Health Education Journal, 72(5), 564-583. https://doi.org/10.1177/0017896912452071.
- [Background] Burki TK. Superbugs: An Arms Race Against Bacteria. Lancet Respir Med. 2018 Sep;6(9):668. doi: 10.1016/S2213-2600(18)30271-6. Epub 2018 Jun 21. No abstract available. PMID 29937248
- [Background] Cave R, Ter-Stepanyan MM, Kotsinyan N, Mkrtchyan HV. An Emerging Lineage of Uropathogenic Extended Spectrum beta-Lactamase Escherichia coli ST127. Microbiol Spectr. 2022 Dec 21;10(6):e0251122. doi: 10.1128/spectrum.02511-22. Epub 2022 Nov 23. PMID 36416548
- [Background] Dadgostar P. Antimicrobial Resistance: Implications and Costs. Infect Drug Resist. 2019 Dec 20;12:3903-3910. doi: 10.2147/IDR.S234610. eCollection 2019. PMID 31908502
- [Background] D'Agata EMC. Addressing the Problem of Multidrug-Resistant Organisms in Dialysis. Clin J Am Soc Nephrol. 2018 Apr 6;13(4):666-668. doi: 10.2215/CJN.13781217. Epub 2018 Mar 22. No abstract available. PMID 29567862
- [Background] Eysenck, M. W., & Keane, M. T. (2015). Cognitive Psychology: A Student's Handbook (7th ed.). Psychology Press. https://doi.org/10.4324/9781315778006.
- [Background] Festinger, L. (1957). A theory of cognitive dissonance (pp. xi, 291). Stanford University Press.
- [Background] Fitria, T. N., Simbolon, N. E., & Afdaleni, A. (2023). Chatbots as online chat conversation in the education sector. International Journal of Computer and Information System (IJCIS), 4(3), 93-104.
- [Background] Hendy A, Al-Sharkawi S, Hassanein SMA, Soliman SM. Effect of educational intervention on nurses' perception and practice of antimicrobial stewardship programs. Am J Infect Control. 2023 Jan;51(1):41-47. doi: 10.1016/j.ajic.2022.05.001. Epub 2022 May 10. PMID 35561943
- [Background] Istepanian RSH. Mobile Health (m-Health) in Retrospect: The Known Unknowns. Int J Environ Res Public Health. 2022 Mar 22;19(7):3747. doi: 10.3390/ijerph19073747. PMID 35409431
- [Background] Kpokiri EE, Ladva M, Dodoo CC, Orman E, Aku TA, Mensah A, Jato J, Mfoafo KA, Folitse I, Hutton-Nyameaye A, Okon-Ben I, Mensah-Kane P, Sarkodie E, Awadzi B, Jani YH. Knowledge, Awareness and Practice with Antimicrobial Stewardship Programmes among Healthcare Providers in a Ghanaian Tertiary Hospital. Antibiotics (Basel). 2021 Dec 22;11(1):6. doi: 10.3390/antibiotics11010006. PMID 35052883
- [Background] Lally, P., van Jaarsveld, C. H., Potts, H. W., & Wardle, J. (2010). How habits are formed: Modelling habit formation in the real world. European Journal of Social Psychology, 40(6), 998-1009.
- [Background] Lawson JH, Niklason LE, Roy-Chaudhury P. Challenges and novel therapies for vascular access in haemodialysis. Nat Rev Nephrol. 2020 Oct;16(10):586-602. doi: 10.1038/s41581-020-0333-2. Epub 2020 Aug 24. PMID 32839580
- [Background] Lutfiyati, H., Thobari, J. A., Yasin, N. M., & Ikawati, Z. (2023). Impact of Educational Programs on the Knowledge and Attitude of Healthcare Professionals in Antimicrobial Stewardship. Indian Journal of Pharmaceutical Education and Research, 57(3), 898-904. https://doi.org/10.5530/ijper.57.3.108.
- [Background] Nezamdoust S, Abdekhoda M, Rahmani A. Determinant factors in adopting mobile health application in healthcare by nurses. BMC Med Inform Decis Mak. 2022 Feb 22;22(1):47. doi: 10.1186/s12911-022-01784-y. PMID 35193552
- [Background] Nguyen, D. B., Arduino, M. J., & Patel, P. R. (2019). Hemodialysis-Associated Infections. Chronic Kidney Disease, Dialysis, and Transplantation, 389-410.e8. https://doi.org/10.1016/B978-0-323-52978-5.00025-2
- [Background] Padigos, J., Ritchie, S., & Lim, A. G. (2020). Enhancing nurses' future role in antimicrobial stewardship. Collegian, 27(5), 487-498. https://doi.org/10.1016/j.colegn.2020.01.005.
- [Background] Pandit R, Awal B, Shrestha SS, Joshi G, Rijal BP, Parajuli NP. Extended-Spectrum beta-Lactamase (ESBL) Genotypes among Multidrug-Resistant Uropathogenic Escherichia coli Clinical Isolates from a Teaching Hospital of Nepal. Interdiscip Perspect Infect Dis. 2020 Apr 15;2020:6525826. doi: 10.1155/2020/6525826. eCollection 2020. PMID 32377184
- [Background] Prestinaci F, Pezzotti P, Pantosti A. Antimicrobial resistance: a global multifaceted phenomenon. Pathog Glob Health. 2015;109(7):309-18. doi: 10.1179/2047773215Y.0000000030. Epub 2015 Sep 7. PMID 26343252
- [Background] Sefah IA, Akwaboah E, Sarkodie E, Godman B, Meyer JC. Evaluation of Healthcare Students' Knowledge on Antibiotic Use, Antimicrobial Resistance and Antimicrobial Stewardship Programs and Associated Factors in a Tertiary University in Ghana: Findings and Implications. Antibiotics (Basel). 2022 Nov 22;11(12):1679. doi: 10.3390/antibiotics11121679. PMID 36551335
- [Background] Vanegas JM, Salazar-Ospina L, Roncancio GE, Jimenez JN. Staphylococcus aureus colonization increases the risk of bacteremia in hemodialysis patients: a molecular epidemiology approach with time-dependent analysis. Am J Infect Control. 2021 Feb;49(2):215-223. doi: 10.1016/j.ajic.2020.05.031. Epub 2020 May 31. PMID 32485274
- [Background] Velazquez-Meza ME, Galarde-Lopez M, Carrillo-Quiroz B, Alpuche-Aranda CM. Antimicrobial resistance: One Health approach. Vet World. 2022 Mar;15(3):743-749. doi: 10.14202/vetworld.2022.743-749. Epub 2022 Mar 28. PMID 35497962
- [Background] WHO. (2019).Thirteenth General Programme of Work, 2019- 2023: Promote health. Keep the world safe Serve the vulnerable. World Health Organization Geneva;.
- [Background] Zong Z, Wu A, Hu B. Infection Control in the Era of Antimicrobial Resistance in China: Progress, Challenges, and Opportunities. Clin Infect Dis. 2020 Dec 23;71(Suppl 4):S372-S378. doi: 10.1093/cid/ciaa1514. PMID 33367579